CLINICAL TRIAL: NCT03225365
Title: Immune Modulation Study in Patients With Metastatic Melanoma Treated With a First Line Therapy of Nivolumab +/- Ipilimumab (IMMUNONIVO/MelpredictPD1).
Brief Title: Nivolumab +/- Ipilimumab Immunomonitoring in Metastatic Melanoma
Acronym: IMMUNONIVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL17_0043
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Nivolumab; Ipilimumab; Immune modulation
MeSH Terms: conditions — Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab (Other): Previous untreated patient with metastatic melanoma eligible for a Nivolumab treatment.
  30 patients will be included in the arm.
  Interventions: Biological: Blood and biopsy sampling
- Nivolumab + Ipilimumab (Other): Previous untreated patient with metastatic melanoma eligible for a Nivolumab + Ipilimumab treatment.
  30 patients will be included in the arm.
  Interventions: Biological: Blood and biopsy sampling

INTERVENTIONS:
Biological: Blood and biopsy sampling — Blood samples (52mL) will be taken at week 1, week 3, week 7, week 13, week 53 or at the progression.
  Skin biopsies will be taken at week 1, week 7, week 53 or at the progression.

SUMMARY:
This is an open bi-centric prospective non-randomized study in patients with metastatic melanoma treated with a first line treatment of Nivolumab +/- Ipilimumab. The aim of the study is to characterize the immune cells modulations under anti-PD-1 +/- anti-CTLA4 and identify the differences between responder and non-responder patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years of age.
* Patient with metastatic or unresectable melanoma
* Nivolumab or Nivolumab + Ipilimumab treatment indication
* Skin biopsies available
* Patient affiliated to or a beneficiary of a social security category.
* Signed Written Informed Consent.
* Patient who agrees to the storage of his biological samples

Exclusion Criteria:

* Treated haematological malignancies Subjects with a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Patients with autoimmune disease.
* Ocular melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change description of biological characteristics of immune cells of the blood by immunomonitoring. | Week 1 (baseline, before the 1st injection), week 3 (before the 2d injection treatment), week 7 (before the 4th) , week 13 (before the 5th), week 53 (before the 26th or during radiological evaluation) or at the progression
  Biological characteristics description of monocytes, dendritic cell and T cells subpopulations including different circulating suppressive subpopulations by immunomonitoring
Change in the immune response by skin biopsy. | Week 1 (Baseline), week 7, week 53 or at the progression.

SECONDARY OUTCOMES:
Progression-free survival | Week1 , every radiological assessments defined by standard care (not by specific time frame)
  Progression free survival (PFS) will be calculated as the period of time from the immunotherapy first administration to the first RECIST 1.1 disease progression
Overall survival | week 1, date of patient death
  Overall survival (OS) will be calculated as the period of time from the immunotherapy first administration to the patient's death.
Auto-immune adverse event frequency | baseline, week 53 or at the progression
  Immune adverse event description by clinical examination and correlation with biological characteristics of immune cells
Subtype of melanoma correlated with biological characteristics of immune cells | baseline
  Subtype of melanoma defined by histological analysis correlated with biological characteristics of immune cells
Immunity gene polymorphism correlated with biological characteristics of immune cells | Week 1, week 3, week 7, week 13, week 53 or at the progression.
  Immunity gene polymorphism defined by RNA sequencing correlated with biological characteristics of immune cells immune cells

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Dermatologie, Centre Hospitalier Lyon Sud (HCL), Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalle S, Verronese E, N'Kodia A, Bardin C, Rodriguez C, Andrieu T, Eberhardt A, Chemin G, Hasan U, Le-Bouar M, Caramel J, Amini-Adle M, Bendriss-Vermare N, Dubois B, Caux C, Menetrier-Caux C. Modulation of blood T cell polyfunctionality and HVEM/BTLA expression are critical determinants of clinical outcome in anti-PD1-treated metastatic melanoma patients. Oncoimmunology. 2024 Jun 26;13(1):2372118. doi: 10.1080/2162402X.2024.2372118. eCollection 2024. PMID 38939518